CLINICAL TRIAL: NCT05246826
Title: The Effect of Conventional Treatment In Addition to Clinical Pilates Exercises in Chronic Neck Pain on Pain Level, Physical, Functional and Psychosocial Status
Brief Title: Comparison of Pilates and Conventional Treatment in Addition to Pilates in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gizem Vaiz Haklıgil, Principal ınvestigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2021-0120
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Chronic Neck Pain
Keywords: pilates; convantional therapy; chronic neck pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pilates Exercises (Experimental): Pilates exercises will be performed 3 days a week, for a total of 18 sessions for 6 weeks.
  Interventions: Other: Clinical Pilates Exercises
- Clinical Pilates Exercises and Conventional Treatment (Experimental): In addition to Pilates exercises, conventional treatment will be performed 3 days a week, for 6 weeks, a total of 18 sessions.
  Interventions: Other: Clinical Pilates Exercises and Conventional Treatment

INTERVENTIONS:
Other: Clinical Pilates Exercises — Pilates exercises; warm-up and cool-down exercises will be performed for 5 repetitions, while other exercises will be performed by the same physiotherapist as 10 repetitions depending on the patient's pain and fatigue. The exercises will be advanced at the end of the 3rd week.
  Arms: Clinical Pilates Exercises
Other: Clinical Pilates Exercises and Conventional Treatment — In addition to pilates exercises, a conventional treatment program will be applied. As part of the conventional treatment program, 20 minutes of Hotpack to the cervical area, 20 minutes of conventional Transcutaneous Electrical Nerve Stimulation (TENS) to the painful area (80 Hertz (Hz), 100 microseconds (μs), until tingling is felt, asymmetrical biphasic rectangular waveform), 8 minutes to the cervical area Ultrasound (US) (4 minutes + 4 minutes, 1.5 watts/cm2, 1 MHz, continuous) will be applied.
  Arms: Clinical Pilates Exercises and Conventional Treatment

SUMMARY:
The aim of this study is to investigate the effects of clinical pilates exercises and electrotherapy on pain level, physical condition, functional status and psychosocial status in patients with chronic neck pain.In the study, individuals will be divided into two groups. Pilates will be applied to one group for 6 weeks, pilates and conventional therapy will be applied to one group. Individuals will be evaluated before and after treatment. In the evaluation, pain, disability, anxiety and depression status, quality of life of individuals will be questioned. In addition, cervical joint range of motion and endurance will be evaluated.

DETAILED DESCRIPTION:
Neck pain is often described by pain and/or stiffness dorsal to the region between the occipital condyles and the C7 vertebra. Pain and/or disability for more than 12 weeks is defined as chronic neck pain. Neck pain is one of the major musculoskeletal disorders in the adult population. Neck pain, which is increasingly prevalent all over the world, significantly affects individuals, families, society, health care systems and businesses. This situation causes serious disability and economic costs. Two-thirds of the entire population faces neck pain at some point in their lives. Its lifetime prevalence ranges from 40% to 70%. The prevalence of neck pain increases with age. It is more common in women approximately in the 5th decade of their life.

In various studies, various changes have been observed in the activation of the superficial and deep neck flexor (DBF) muscles of individuals experiencing neck pain. In studies conducted with electroneuromyography, it was determined that neuromuscular muscle activation increased more in superficial muscles, and decreased undesirably in DBF muscles. DBF muscles provide a fundamental contribution to the preservation of physiological cervical lordosis and the maintenance of spine stability in cranio-vertebral junction movements. For this reason, exercise methods for gaining strength and endurance of these muscles have become very important recently.

The neck region contains deep suboccipital muscles with dense muscle spindles, nerve connections to the vestibular and visual systems. Especially the high muscle spindle density in the superior and inferior oblique muscles and the rectus capitis posterior major and minor muscles is important in terms of proprioceptive input in coordinated head-eye movements. In a disorder in the neck region, muscle dysfunction occurs as a result of pain, disruption of sensory-motor input, and the transfer of deep muscles to superficial muscles. All these problems can cause asymmetrical, tight, position and movement of the neck to be perceived abnormally.

Fear avoidance beliefs are significantly associated with the experience of pain, especially when the pain becomes chronic. The anticipated threat of intense pain often causes constant alertness of pain dermatomes. This can cause even low-intensity pain sensations to be unbearable for the person. Only the increased expectation of pain or re-injury can further encourage avoidance behaviors. Increased pain or fear of re-injury interferes with many activities. Studies have shown that fear of movement in chronic neck pain increases pain and disability, worsens functional status, and negatively affects physical performance.

Studies associate individuals who experience persistent neck pain with psychological factors, including cognitive stress, anxiety, and depressed mood. In addition, it has been reported that sleep disorders are seen in parallel with the severity of pain in patients with chronic neck pain. These psychological factors may play a role in the chronicity of symptoms and cause increased pain, disability or fear-avoidance.

Studies have shown that chronic neck pain is associated with low quality of life. It has been stated that the quality of life of patients with chronic neck pain is worse than normal individuals, and that many of these individuals face mental problems and may also experience psychosocial disorders such as anxiety and depression.

Clinical Pilates exercises are a set of exercises that emphasize mind-body unity. Pilates strengthens the deep stabilizing muscles of the spine, gives flexibility to the spine, develops mind-body awareness and improves posture. Pilates also promotes the activation of the deep neck flexor muscles by promoting a neutral position of the cervical spine with mild upper cervical flexion at the cranio-cervical junction. Studies investigating the effect of clinical pilates on pain and disability in patients with chronic neck pain have shown that clinical pilates is effective in these parameters. Although it has been shown that neck perception is associated with factors such as pain, disability, anxiety and quality of life, no study has been found in the literature examining the effects of exercise and electrotherapy methods on neck awareness. In addition, there was no study examining the effect of electrotherapy on fear of movement and fear avoidance beliefs in individuals with chronic neck pain, and the effects of clinical pilates exercises on body awareness, fear of movement, and biopsychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Individuals with neck pain lasting longer than 3 months
* Individuals with a score of 3 or more according to VAS

Exclusion Criteria:

* Those with a history of surgery
* Those who have received physical therapy for the neck region in the last 6 months
* With pregnancy status
* Cancer, infectious disease
* With inflammatory disease
* With neurological disease
* Joint injection in the last 3 months
* Individuals using analgesics, myorelaxants, or antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 6 weeks
  Pain intensity will be evaluated by VAS. Individuals are asked to mark the intensity of pain. felt on a 10-centimeter horizontal line. The score obtained by measuring with a tape measure will be used in the analysis. High scores are associated with increased pain. 0 means no pain, 10 means untolerable pain.

SECONDARY OUTCOMES:
Cervical Normal Joint Movement | 6 weeks
  Cervical flexion, extension, lateral flexion (right-left), rotation (right-left), normal joint motion will be actively evaluated with a goniometer in 2 repetitions and the best score will be recorded in degrees for the analysis . Grades close to the normal joint range of motion criteria indicate that the individual has a good range of motion.
Cervical Flexor Muscle Endurance Test | 6 weeks
  Neck Flexor Muscle Endurance Test: Individuals will be asked to take the chin-tuck position while in the supine hook position. Afterwards, he will be asked to maintain his position by raising his head 2.5 cm above the ground. The time during which the head position is maintained will be recorded in seconds.
Cervikal Extensor Muscle Endurance Test | 6 weeks
  Neck Extensor Muscle Endurance Test: Individuals will be asked to lie face down with the head ahead of the bed and keep the head horizontal. The time during which the jaw retraction and head position can be maintained will be recorded in seconds. The test will be stopped when the test loses its position and feels unbearable pain.
Strength and Endurance of Deep Cervical Flexors | 6 weeks
  Deep flexor muscle strength and endurance will be assessed using the craniocervical flexion test. The test is performed with a biofeedback pressure unit (Stabilizer Pressure Biofeedback-Chattanooga Stabilizer). Subjects are asked to lie on their back with their head in a neutral position and knees bent. The pressure unit is placed in the suboccipital region. The unit is inflated to 20 mmHg of mercury. The person is asked to do 10 contractions lasting 10 seconds at 5 different pressure levels (22,24,26,28,30). Performance index and Activation score will be calculated to be used in the analysis.
Functional Status-Neck Disability Index | 6 weeks
  Neck Disability Index: It will be used to evaluate disability. It includes 10 questions, 7 about activities of daily living, 2 questions about pain and 1 question about concentration. Each question is evaluated with 6 response options that can be scored between 0 (no pain and limitation) and 5 (maximum pain and limitation).The total score ranges from 0 to 50, and higher scores indicate more limitations.
Functional Status-Fremantle Neck Awareness Questionnaire: | 6 weeks
  Fremantle Neck Awareness Questionnaire: Likert-type assessing individual-specific altered perception (0 = Never/Never feel this way, 1 = I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I feel this way often, 4 = Always or this is how I feel most of the time) is a simple survey. The questionnaire asks individuals 9 questions such as how they perceive their neck relative to their body, how they perceive their body position.Higher scores indicate decreased awareness.
Psychosocial Factors-Neckpix Scale: | 6 weeks
  It was developed to evaluate the fear of movement in patients with chronic neck pain. In the scale, activities of daily living for neck pain are shown with 10 different pictures. The fear of movement experienced during activities will be asked to evaluate between 0-10 points. The total score is 100 and 100 means greatest fear
Psychosocial Factors-Fear Avoidance Beliefs Questionnaire (KKIA) | 6 weeks
  It consists of 16 questions and 2 parts. In the first part, there are physical activities, in the second part there are questions about work. In the questionnaire, which is evaluated with a 7-point Likert type scale, physical activities are scored between 0-24, while questions about work are scored between 0-36. A high score indicates that the person has high fear avoidance beliefs.
Psychosocial Factors-Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  It is used to reveal the anxiety and depression accompanying the existing diseases in the individual. The scale consists of two subscales and 14 questions. 7 questions consisting of odd numbers evaluate anxiety (HADS-A), and 7 questions consisting of even numbers evaluate depression (HADS-D). Each question has 4 answer options that can be answered between 0-3 points. For both sub-scales; A score of 0-7 is considered 'normal', a score of 8-10 a 'probable case', and a score of 11-21 a 'probable case of anxiety/depression
Psychosocial Factors-Cognitive Exercise Therapy Method Scale (BETY Scale) | 6 weeks
  The scale consists of 30 items and a 5-point Likert system is used to calculate the scores. For each item, there are 4 response options that can be scored between 0 (No/never) and 4 (Yes/always). The total score is given over 30 items, and high scores indicate that the biopsychosocial status of the individual is adversely affected
Quality of Life-Short form -36 | 6 weeks
  the quality of life of individuals will be evaluated with the Short Form-36. The questionnaire evaluates the perception of individuals' general health, social and physical functions, vitality, mental health, role limitations and pain due to physical and emotional problems, with a total of 11 questions and 36 items under 8 sub-titles. Each title is calculated separately and points are given between 0-100.The subscales are scored between 0-100 and higher scores reflect better
Patient Satisfaction | 6 weeks
  On a 10 cm long line to determine their satisfaction level after the treatment; It will be asked to mark with a pencil by grading from 0 (not at all satisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: SEVİM ÖKSÜZ, Asst. Prof., Study Director — Eastern Mediterranean University; Ender Angın, Assoc. Prof., Study Director — Eastern Mediterranean University
Locations (1):
- Gizem Vaiz Haklıgil, Famagusta, Cyprus